CLINICAL TRIAL: NCT05360199
Title: Are Postoperative Patient Patient Reported Outcome Measures Influenced by Recall of Preoperative Scores? - a Randomized Controlled Trial
Brief Title: Are Postoperative Patient PROMS Influenced by Recall of Preoperative Scores?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Principal Investigator, Pedro Daniel Valente Aguiar, Doctor, Centro Hospitalar De São João, E.P.E.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHSJ1989
Record Dates: First submitted 2022-04-23; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Degenerative Diseases, Spinal Cord
Keywords: PROM; Recall bias
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: patients are unaware whether they are in the intervention or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): no recall PROMs group ; without knowledge of previous PROMs scores
- intervention group (Active Comparator): recall PROMs group ; with knowledge of previous PROMs scores
  Interventions: Behavioral: PROMs

INTERVENTIONS:
Behavioral: PROMs — evaluate the impact of recall bias on post proms scores
  Arms: intervention group

SUMMARY:
To evaluate whether postoperative PROM scores of spine patients are influenced by memory bias

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with valid preoperative PROM scores submitted to spine surgery due to degenerative pathology from January 2019 to April 2020 at our center (spine unit of a neurosurgical department in a Portuguese university hospital) were included in the study and received PROMs questionnaires with a letter of consent.

Exclusion Criteria:

* Patients without valid preoperative questionnaires were excluded from the study while patients were lost to follow-up if mail questionnaires were not completed two months after PROMs remittance or if they had submitted incomplete or invalid answers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Median COMI score results | 4 weeks
  Core outcome measures index. Scale 0 to 10 where 0 means the best score

SECONDARY OUTCOMES:
Median ODI score | 4 weeks
  Neck disability index Oswestry disability index. Scale 0 to 100 where 0 means the worst score
Median EQ-5D score | 4 weeks
  EuroQol 5 D where 1 is the best score and -0,500 the worst score
Median NDI | 4 weeks
  Neck disability index Scale 0 to 100 where 0 means the worst score

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Centro Hospitalar Universitário São João, Porto
  - Centro Hospitalar Universitário São João, Portugal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT05360199/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT05360199/SAP_001.pdf